CLINICAL TRIAL: NCT03660332
Title: The Effect of an Acute Increase in Plasma IL-6 on Glucose Tolerance When a Meal is Administered Intraduodenally
Acronym: DUIL-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Lang Lehrskov, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-16036538
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Postprandial Glucose Homeostasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-6 infusion (Active Comparator): Healthy young men will receive IL-6 infusion
  Interventions: Procedure: Infusion of a liquid meal intraduodenally
- Placebo infusion (Placebo Comparator): Healthy young men will receive saline infusion
  Interventions: Procedure: Infusion of a liquid meal intraduodenally

INTERVENTIONS:
Procedure: Infusion of a liquid meal intraduodenally — Infusion of IL-6/NaCL before a liquid meal intraduodenally

SUMMARY:
The aim of the study is to investigate and clarify whether the effect of IL-6 on glucose tolerance and insulin secretion are secondary to the changes in gastric emptying.

The literature provides no information regarding a role for interleukin-6 (IL-6) in the regulation of beta cell function (glucose or meal-stimulated insulin secretion) in humans. Previous studies infusing IL-6 into humans have primarily focused on insulin action and the effects on peripheral insulin sensitivity whereas a potential effect on insulin secretion has been neglected.

We have demonstrated that an acute increase in IL-6, obtained by a single bolus of IL-6, potentiated glucose-induced insulin secretion in a glucagon-like peptide-1 (GLP-1) dependent manner in mice1. In mice, IL-6 enhanced insulin secretion in a dose- and glucose-dependent manner, along with increasing concentrations of GLP-1. Interleukin-6 had no effect on insulin secretion in GLP-1 receptor knock-out mice or in mice treated with the GLP-1 receptor antagonist. Thus, in mice, GLP-1 has proven an essential mediator of IL-6 actions on beta cell function.

Importantly, a single bolus of IL-6 also significantly increased glucose-stimulated insulin secretion in several mouse models of obesity and diabetes (diet-induced obesity, the ob/ob and the db/db mouse).

Own data show that an infusion of IL-6 causes a significant delay in the rate of gastric emptying (GE) after a mixed meal in healthy young men. Data showed that this delay in GE is associated with much improved glucose tolerance and insulin secretion (unpublished data).

In the present study we wish to investigate whether the beneficial effects of IL-6 on postprandial glucose tolerance and insulin secretion are dependent on a delay in gastric emptying. We will bypass the ventricle and infuse a mixed meal directly into the duodenum of healthy young men.

This study has the potential to show that the known effect of IL-6 on postprandial glucose tolerance is dependent on a delayed GE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 35 years
* Healthy (based on screening)

Exclusion Criteria:

* Smoking
* BMI < 18 and > 25 kg/m2
* Evidence of severe thyroid, liver, lung, heart or kidney disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
The paracetamol uptake | 0-14 days
  paracetamol blood levels (mmol/l) on both study days. The paracetamol absorbance will be compared between the 2 study days.

SECONDARY OUTCOMES:
GLP-1 secretion | 0-14 days
  Active GLP-1 blood levels on both study days. The levels on the 2 study days will be compared.
Glucagon secretion | 0-14 days
  Glucagon blood levels on both study days. The levels on the 2 study days will be compared.
Insulin levels | 0-14
  Insulin blood levels on both study days. The levels on the 2 study days will be compared.
Glucose | 0-14
  Plasma glucose levels on both study days. The levels on the 2 study days will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Professor, Study Director — CFAS, Rigshospitalet
Locations (1):
- Rigshospitalet, Centre of Inflammation and Metabolism (CIM) Centre for Physical Activity Research (CFAS), Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lang Lehrskov L, Lyngbaek MP, Soederlund L, Legaard GE, Ehses JA, Heywood SE, Wewer Albrechtsen NJ, Holst JJ, Karstoft K, Pedersen BK, Ellingsgaard H. Interleukin-6 Delays Gastric Emptying in Humans with Direct Effects on Glycemic Control. Cell Metab. 2018 Jun 5;27(6):1201-1211.e3. doi: 10.1016/j.cmet.2018.04.008. Epub 2018 May 3. PMID 29731416